CLINICAL TRIAL: NCT05066204
Title: Evaluation of Different Teaching- and Learningmethods Concerning the Humeral Intraosseal Access in Inexperienced Providers
Brief Title: Evaluation of Different Teaching- and Learningmethods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Thomas Ott, Thomas Ott, M.D., DESA, Scientific consultant of the simulation center, Department of Anesthesiology, University Hospital Center, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021-16112 EK RLP
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Complication of Infusion; Education, Medical

STUDY DESIGN:
Intervention Model Description: Two unbound samples running through a different sequence of teching-/learningmethods
Who Masked: Investigator
Masking Description: Investigator are blinded/masked against the study arm of the particular assessed participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence: self-study, then teaching video (Other): Participants first do self-study, then right afterwards watch a teaching video, then become tested on a simulator and are videorecorded for evaluation
  Interventions: Other: Sequence of teaching-/learningmethod
- Sequence: teaching video, then self study (Other): Participants first watch a teaching video, then do self-study, then become tested on a simulator and are videorecorded for evaluation
  Interventions: Other: Sequence of teaching-/learningmethod

INTERVENTIONS:
Other: Sequence of teaching-/learningmethod — see: arm/group descriptions

SUMMARY:
Due to the corona pandemia and the consecutive reduction of teaching students face to face the imparting of medical skills is limited. Video sequences may be an adequate alternative to educate selected practical skills. The investigators explored this aspect in spring 2021 concerning the humeral intraosseous access. This study was registered under ClinicalTrials: NCT04842357. Data is still under statistical analysis and not published yet. As a secondary endpoint we found participant having done self-study first and watched a teaching-video one week later performed better than participant in the vice versa sequence. This may have important curricular implications. So, we launch the present study to investigate, if the sequence: Self-Study, then Teaching-Video is more efficient than vice versa.

DETAILED DESCRIPTION:
The investigators will recruit last year medical students and randomise them into two groups: Group A and Group B. Group A will watch a standardised video about the skill, then directly do self-study. Group B will do self-study and then directly watch a standardised video. Right after this, both groups will be video recorded during the performance of the skill: humeral intraosseous access on a simulator. The performance will be quantified by a scale by two investigators

ELIGIBILITY:
Inclusion Criteria:

* voluteer medical students in their last year of medical school (i.e. after 2nd state board in Germany)
* writen informed consert

Exclusion Criteria:

* denial of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
sum of score | 1 Day
  sum of the score used to evaluate the particpants' performance by video records

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Centre Mainz, Mainz, RLP, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ott T, Demare T, Mohrke J, Silber S, Schwab J, Reuter L, Westhphal R, Schmidtmann I, Dietz SO, Pirlich N, Ziebart A, Engelhard K. Does an instructional video as a stand-alone tool promote the acquisition of practical clinical skills? A randomised simulation research trial of skills acquisition and short-term retention. BMC Med Educ. 2024 Jul 2;24(1):714. doi: 10.1186/s12909-024-05714-6. PMID 38956562